CLINICAL TRIAL: NCT05455164
Title: The Effect of Eucaloric High-Protein Fiber Diet on Anthropometric and Metabolic Profile of Healthy Adults: A Repeated Single-Arm Clinical Trial
Brief Title: The Effect of Eucaloric High-Protein Fiber Diet in Healthy Adults: A Repeated Single-Arm Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Katolik Widya Mandala Surabaya (Other)
Responsible Party: Principal Investigator, Hendy Wijaya, Head of Clinical Pharmacology research laboratories, Universitas Katolik Widya Mandala Surabaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0295/WM12/KEPK/DSN/T/2022
Record Dates: First submitted 2022-07-05; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Dietary Exposure
Keywords: isomalto-oligosaccharide; blood glucose; cholesterol; fibre diet

STUDY DESIGN:
Intervention Model Description: A Repeated Single-Arm Clinical Trial The aims of this study is to investigate the effect of eucaloric high protein and fiber diet on healthy subjects. Thirteen healthy subjects, age 29,85 ± 4,06 years old, with body mass index (BMI) 29,55 ± 4,12 kg/m2 were prescribed eucaloric high protein diet for two weeks, followed by washing period for two week. Then, they were prescribed with eucaloric high protein and high fiber diet for two more weeks. Twenty grams of dietary fiber were in the form of isomaltooligosaccharides (IMO) based creamer formulae. Their body composition, waist circumference, fasting blood glucose, blood uric acid and total cholesterol concentration were measured after every dietary intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Without supplementation, followed by Supplementation with Dietary Fibre (Other): For the first two weeks, subjects were given eucaloric prepared meals typical of Indonesian diet, which has low protein and low DF contents (contain less than 15 g/d of DF and protein content less than 15% of total macronutrient distribution range).
  After two weeks of washing periods, all of the subjects were given eucaloric prepared meal which contain high protein and DF (contain 25-30 gram DF and protein content between 30-40% of total macronutrient distribution range). At the end of interventions, waist circumference, body weight, body composition, fasting plasma glucose, uric acid, and total cholesterol were measured again. Half of DF content in food came from natural occurring fiber from fruit, vegetables and whole grains, the other half (50%) come from IMO-based fiber supplement (FibercremeⓇ, PT. Lautan Natural Krimerindo, Mojokerto, Indonesia
  Interventions: Dietary Supplement: Isomalto Oligosaccharide

INTERVENTIONS:
Dietary Supplement: Isomalto Oligosaccharide — all of the subjects were given eucaloric prepared meal which contain high protein and DF (contain 25-30 gram DF and protein content between 30-40% of total macronutrient distribution range)

SUMMARY:
The aims of this study is to investigate the effect of eucaloric high protein and fiber diet on healthy subjects.

DETAILED DESCRIPTION:
Several studies have shown that high protein diet can reduce body fat, increase muscle mass, and improve some metabolic parameters of subjects. Also, several studies have shown that high intake of fiber could reduce body weight and improve cardiometabolic parameters. Therefore, combining high-protein diet and high-fiber diet should have a positive synergistic effect on several of anthropometric and metabolic parameters. The aims of this study is to investigate the effect of eucaloric high protein and fiber diet on healthy subjects. Thirteen healthy subjects, age 29,85 ± 4,06 years old, with body mass index (BMI) 29,55 ± 4,12 kg/m2 were prescribed eucaloric high protein diet for two weeks, followed by washing period for two week. Then, they were prescribed with eucaloric high protein and high fiber diet for two more weeks. Twenty grams of dietary fiber were in the form of isomaltooligosaccharides (IMO) based creamer formulae. Their body composition, waist circumference, fasting blood glucose, blood uric acid and total cholesterol concentration were measured after every dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* (BMI) of >= 25.0
* Healthy subjects

Exclusion Criteria:

* pregnant,
* under any medication
* having any kind of diseases and acute infection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
body composition analysis (Arm-, Trunk-, Leg Fat composition) | 2 weeks after meal
  in Kg or %
Fasting Plasma Glucose | 2 weeks after meal
  Fasting Plasma Glucose mmol/dl
Plasma Uric Acid | 2 weeks after meal
  Plasma Uric Acid mg/dl
Total Cholesterol | 2 weeks after meal
  Total Cholesterol Mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Hendy Wijaya, MD.M.Biomed., Principal Investigator — Faculty of Pharmacy, Universitas Katolik Widya Mandala Surabaya
Locations (1):
- Universitas Katolik Widya Mandala Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided